CLINICAL TRIAL: NCT05889351
Title: A Phase IIa, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of 3% LTX-109 Compared to Placebo for Nasal Decolonisation of Staphylococcus Aureus.
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of 3% LTX-109 for Nasal Decolonisation of Staphylococcus Aureus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharma Holdings AS (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C22-109-08
Record Dates: First submitted 2023-05-02; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Nasal Decolonization of Staphylococcus Aureus
MeSH Terms: interventions — L-arginyl-2,5,7-tris(1,1-dimethylethyl)-L-tryptophyl-N-(2-phenylethyl)-L-argininamide; Gels

STUDY DESIGN:
Intervention Model Description: Randomised, Double-blind, Placebo-controlled Randomization 2:1, active to placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Vehicle treatment
  Interventions: Drug: Vehicle gel, 4 + 4 applications or 4 + 2 applications
- Cohort 1 (Active Comparator): For all subjects, the IMP was applied 4 times during an intensive dosing regimen for 4 ½-hours (on Day 1 at 0, 1 ½, 3 and 4 ½ - hours). For subjects in Cohort 1, this was followed by 4 additional applications: on Day 1 at 12 hours, on Day 2 at 24 and 36 hours, and on Day 3 at 48 hours.
  Interventions: Drug: LTX-109 3% gel, 4 + 4 applications
- Cohort 2 (Active Comparator): For all subjects, the IMP was applied 4 times during an intensive dosing regimen for 4 ½-hours (on Day 1 at 0, 1 ½, 3 and 4 ½ - hours). For subjects in Cohort 2 the IMP was likewise applied 4 times during the 4 ½-hour period (on Day 1 at 0, 1 ½, 3 and 4½ hours), but was followed by 2 applications: on Day 1 at 12 hours and on Day 2 at 36 hours.
  Interventions: Drug: LTX-109 3% gel, 4 + 2 applications

INTERVENTIONS:
Drug: Vehicle gel, 4 + 4 applications or 4 + 2 applications — Control arm/placebo
  Arms: Placebo
Drug: LTX-109 3% gel, 4 + 4 applications — Cohort 1 active treatment
  Arms: Cohort 1
Drug: LTX-109 3% gel, 4 + 2 applications — Cohort 2 active treatment
  Arms: Cohort 2

SUMMARY:
A Phase IIa, double-blind, placebo-controlled, randomised study designed to evaluate the efficacy, safety and tolerability of two dosing regimens with LTX-109 administered topically to the anterior nares in subjects with persistent carriage of Staphylococcus aureus (S. aureus).

DETAILED DESCRIPTION:
Approximately 90 subjects planned screened to achieve 27 randomised and dosed subjects with persistent S. aureus carriage.

On Day 1, subject randomisation in a 2:1 ratio to receive either LTX-109 (n=18) or placebo (n=9). Cohort (1 [8 doses] or 2 [6 doses]) used as a stratification variable to preserve the 2:1 treatment randomisation ratio in each cohort (LTX-109 n=9 or placebo n=5/4).

For all subjects, the IMP was to be applied 4 times during an intensive dosing regimen for 4 ½-hours (on Day 1 at 0, 1 ½, 3 and 4 ½ - hours). For subjects in Cohort 1, this was followed by 4 additional applications: on Day 1 at 12 hours, on Day 2 at 24 and 36 hours, and on Day 3 at 48 hours. For subjects in Cohort 2 the IMP was likewise applied 4 times during the 4 ½-hour period (on Day 1 at 0, 1 ½, 3 and 4½ hours), but was followed by 2 applications: on Day 1 at 12 hours and on Day 2 at 36 hours. On each dosing occasion, a large drop (approximately 250 μL) of IMP was applied into each nostril and distributed to cover the whole area of the nostril. The subjects were carefully monitored by clinical staff during and after dosing. Safety assessments (AEs, vital signs, safety laboratory assessments and local tolerability) and efficacy assessments (nasal swab) were performed.

All subjects were instructed to wash the body and hair with chlorhexidine body wash and shampoo at the CRU on Day 1 (prior to the first dose) and on Day 2. Subjects were provided with chlorhexidine body wash and shampoo for body and hair wash at home on Day 3, Day 4, Day 5, Day 6 and Day 7. On Day 3 and Day 7, subjects used the chlorhexidine shower before the visits to the CRU.

A final end-of-study visit (Visit 5) took place on Day 7 (+2 days) or after early withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the study.
* Male or female subject aged 18 to 65 years, inclusive.
* Persistent nasal carrier of S. aureus (MSSA), confirmed by 2 positive bacterial cultures from the nose during the screening period.
* Medically healthy subjects without abnormal clinically significant medical history, physical findings, vital signs, or laboratory values at the time of screening, as judged by the Investigator.
* Women of child bearing potential (WOCBP) had to practice abstinence (only allowed when this was the preferred and usual lifestyle of the subject) or had to agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy from the date of dosing until 2 weeks after last dose. Female subjects had to refrain from donating eggs from the date of dosing until 3 months after dosing with the IMP. Their male partner had to agree to use a condom from date of first dosing until 2 weeks after last dose if he had not undergone vasectomy.

Male subjects had to be willing to use condom or had to be vasectomised or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and had to refrain from donating sperm from the date of dosing until 3 months after dosing with the IMP. Their female partner of child-bearing potential had to use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above).

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, could either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the administration of IMP.
* Severe eczema or skin wounds, dry or sensitive skin assessed as clinically significant by the Investigator.
* Any positive result at screening for serum hepatitis B surface antigen, hepatitis C antibody and HIV.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to LTX-109 or chlorhexidine.
* S. aureus (MSSA and/or MRSA) decolonisation attempt in the 6 months prior to - MRSA positive at screening (Visit 1 and/or Visit 2).
* Inability to take medications nasally.
* Nasal polyps or significant anatomical nasal abnormality, as judged by the Investigator.
* Evidence of open wound, lesion, inflammation, erythema or infection (including active rhinitis, sinusitis or upper respiratory infection or severe acne vulgaris) affecting the nostril area, lip and skin close to the nose.
* History of multiple episodes (>3) of epistaxis within 12 months prior to screening Visit 2.
* Disease in the region of the application sites, significant history of trauma or skin disease in the region of the application sites, current nasal skin or nasal septum condition requiring treatment or nasal surgery in the 6 months prior to screening Visit 2.
* In situ nasal jewellery or open nasal piercings.
* Previous or concurrent treatment with antimicrobials for an infection within the last 28 days prior to the first administration of IMP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Operating Window Eradication | 6 hour to 12 hours after start of treatment
  Number of subjects on LTX-109 versus placebo with bacterial eradication period lasting for 6 hours, from 6 to 12 hours after start of treatment (the "Operation Window").

SECONDARY OUTCOMES:
Number eradicated at specific timepoints | 4.5 hours, 6 hours, 12 hours
  Number of subjects on LTX-109 versus placebo with bacterial eradication at 4 ½, 6 and 12 hours after start of treatment.
Percentage change in colony forming units (CFUs) in subjects from baseline | 4.5 hours, 6 hours, 12 hours
  Percentage change in colony forming units (CFUs) in subjects from baseline on LTX-109 versus placebo at 4 ½, 6 and 12 hours after start of treatment.
Number of subjects on LTX-109 versus placebo with bacterial eradication period lasting for 48 hours | From 6 hours to 54 hours after start of treatment
  Number of subjects on LTX-109 versus placebo with bacterial eradication period lasting for 48 hours, from 6 to 54 hours after start of treatment ("48 hours Eradication Window")
Adverse events | Through treatment and followup of 7 days
  Occurrence and frequency of adverse events (AEs)
Local tolerability assessed by health care professional | Pre-dose, 1.5 hours, 4.5 hours, 6 hours, 12, hrs, 54 hours and Day 7
  Incidence of local reactions (erythema, swelling and lesions) will be assessed. Each nostril will be evaluated separately and each parameter will be scored using a 4-graded scale (0-3): 0: none,1: mild, 2: moderate, 3: severe
Local tolerability assessed by the subject | Pre-dose, 1.5 hours, 4.5 hours, 6 hours, 12, hrs, 54 hours and Day 7
  Incidence of local reactions (pruritus and discomfort) will be assessed by the subject. Each nostril will be evaluated separately using a visual analogue scale (VAS).
Asessment of Vital Signs (Systolic and diastolic blood pressure and pulse) | 24 hours, 54 hours and Day 7
  Systolic and diastolic blood pressure (BP) and pulse will be measured in supine position after 10 minutes of rest
Safety laboratory assessments | 54 hours and Day 7
  Blood samples for the analysis of clinical chemistry and haematology be collected through venepuncture or an indwelling venous catheter and sent to the certified clinical chemistry laboratory and analysed by routine analytical methods. Safety laboratory values will be specified and documented as normal, abnormal NCS, or abnormal CS in the eCRF. Abnormal values assessed by the Investigator as CS will be reported as AEs. Clinical chemistry parameters to be reported: Alanine aminotransferase (ALT),Albumin, Alkaline, phosphatase (ALP), Aspartate aminotransferase (AST), Bilirubin (total and conjugated), Calcium, Creatinine (eGFR included), Glucose, Phosphate, Potassium, Sodium, Urea. Haematology parameters to be reported: Red blood cell (RBC) count, White blood cell (WBC) count with differential count, Haematocrit (B-EVF), Haemoglobin (Hb), Platelet count.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Nilsson, MD, Phd, Principal Investigator — ClinSmart AB
Locations (1):
- ClinSmart Sweden AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No